CLINICAL TRIAL: NCT02589353
Title: The Role of Salivary Contents in Taste Perception of Starch and Its Hydrolysis Products
Brief Title: Human Oral Detection of Glucose Olygomers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Juyun Lim, Associate Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB # 5373
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Acarbose

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acarbose (Experimental): Acarbose solution will be swabbed on the tip of the tongue to inhibit salivary alpha amylase activity; each swab will contain ~484 microgram acarbose; total maximum exposure of each subject to acarbose will be ~14-30 mg each session (1-20 sessions)
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Acarbose — Acarbose solution will be swabbed on the tip of the tongue to inhibit salivary alpha amylase activity; each swab will contain ~484 microgram acarbose; total maximum exposure of each subject to acarbose will be ~14-30 mg each session (1-20 sessions)

SUMMARY:
Although salivary contents play a major role in the early stage of food digestion process, their role in taste perception of glucose polymers is essentially unknown. It is hypothesized that the differences in salivary contents, more specifically salivary amylase concentration and activity, influence taste perception of glucose polymers and ultimately eating behavior, which is related to risks in various diseases. The current project will investigate the variation in salivary contents across individuals and its role in taste perception of glucose polymers.

ELIGIBILITY:
Inclusion Criteria:

* self-reported healthy adults between the ages of 18-60 who are fluent in English.

Exclusion Criteria:

* adults 61 years old and above
* smokers
* pregnant women
* taking any prescription pain/ insulin medication
* has a history of taste or smell loss or other oral disorders (e.g., burning mouth syndrome)
* has current oral lesions, canker sores, or piercings
* has a history of food allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Detection of glucose polymers in the presence of acarbose | up to 5 years
  There is only one outcome measure, that is the detection of glucose polymers. Subjects will be asked to discriminate a target sample (glucose polymers). Three samples will be applied using cotton swabs on the subjects' tongue (one at a time): 2 blanks (water + acarbose) and 1 target stimuli (glucose polymer solution + acarbose). Subjects will be asked to identify the target sample. The number of subjects who correctly identify the target stimuli will be counted and will be statistically analyzed to determine whether glucose polymer can be detected without the confounding effect of salivary alpha amylase hydrolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Juyun Lim, Principal Investigator — Oregon State University
Locations (1):
- Department of Food Science and Technology, Corvallis, Oregon, United States